CLINICAL TRIAL: NCT04446091
Title: A Clinical Study of Exploring Camrelizumab in the Treatment of Colorectal Mucinous Adenocarcinoma(MAC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChiECRCT20200108
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal mucinous adenocarcinoma (MAC),Camrelizumab,PD-1,anti-angiogenic drugs
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-drug group (Experimental): Camrelizumab:200mg,iv,Q2W; Fruquintinib:5mg,po.qd,Day1~21, repeat every 28 days;or Regorafenib: 80mg,po.qd,Day1~21, repeat every 28 days;or Apatinib:250mg,po.qd,Day1~21, repeat every 28 days;
  Interventions: Drug: Carilizumab + anti-angiogenic TKIs (available with fuquitinib, rigofenib, apatinib, etc.)
- Three-drug group (Experimental): Camrelizumab:200mg,iv,Q3W; Irinotecan:150mg/m2,iv 30~90min,d1,Q3W Fruquintinib:5mg,po.qd,Day1~21, repeat every 28 days;or Regorafenib: 80mg,po.qd,Day1~21, repeat every 28 days;or Apatinib:250mg,po.qd,Day1~21, repeat every 28 days;
  Interventions: Drug: Carilizumab + anti-angiogenic TKIs (available with fuquitinib, rigofenib, apatinib, etc.)+Irinotecan

INTERVENTIONS:
Drug: Carilizumab + anti-angiogenic TKIs (available with fuquitinib, rigofenib, apatinib, etc.) — Observe the efficacy of immune checkpoint inhibitors combined with anti-angiogenic drugs for colorectal mucinous adenocarcinoma
  Arms: Two-drug group
Drug: Carilizumab + anti-angiogenic TKIs (available with fuquitinib, rigofenib, apatinib, etc.)+Irinotecan — Observe the efficacy of immune checkpoint inhibitors combined with anti-angiogenic drugs and chemotherapy for colorectal mucinous adenocarcinoma
  Arms: Three-drug group

SUMMARY:
This is an open-label, single center, non-randomized, phase Ⅱ trial to evaluate safety and efficacy of using the combination treatment of Camrelizumab with anti-angiogenic drugs and Chemotherapy of metastatic colorectal mucinous adenocarcinoma(MAC).

DETAILED DESCRIPTION:
Colorectal cancer contains multiple pathological types, and one of the more special pathological types is mucinous adenocarcinoma. The prognosis of patients with mucinous adenocarcinoma is not ideal.Some molecular and genetic factors may be related to the characteristics of mucinous adenocarcinoma, in which microsatellite instability and loss of mismatch repair proteins are a focus of current research. Microsatellite instability is often associated with poor differentiation and higher tumor stage. Adenocarcinoma that secretes a large amount of mucus in pathological features.so,In this study, the incidence of ORR and AEs was the main endpoint, and the efficacy and safety of Camrelizumab combined with anti-angiogenic drugs in the treatment of advanced colorectal mucinous adenocarcinoma were observed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Join the study voluntarily and sign the informed consent;
* 2. Unresectable locally advanced or metastatic colorectal mucinous adenocarcinoma or colorectal adenocarcinoma containing mucinous gland components diagnosed by histopathology or cytology;
* 3. Patients who have received at least first-line and above systemic chemotherapy (which may include platinum, fluorouracil, or irinotecan-based) progress or intolerance (maintenance treatment progress after first-line chemotherapy can also be included). Simultaneous chemoradiotherapy for recurrence or metastasis after surgery is considered as first-line treatment; for radical concurrent chemoradiotherapy, neoadjuvant/adjuvant therapy (chemotherapy or radiochemotherapy), if disease progression occurs during treatment or within 6 months after stopping treatment, It should be counted as a failure of first-line treatment;
* 4. Age 18-75 years old (including boundary value, calculated on the day of signing informed consent), both men and women;
* 5. ECOG score 0-2 points;
* 6. Blood routine and liver and kidney function meet the following conditions: neutrophil count>1.5*10^9/L, hemoglobin concentration>90g/L, platelet count>80*109/L; ALT and AST<2.0*ULN (with liver The transferee may be <5.0*ULN);
* 7. Estimated survival time> 3 months;
* 8. Willing to accept long-term follow-up, willing to provide tumor tissue samples, willing to provide blood samples before and after treatment;

Exclusion Criteria:

* 1. Known predisposition of inherited or acquired bleeding and thrombosis (such as hemophiliacs, coagulopathy, thrombocytopenia, etc.);
* 2. Urinary routines suggest that urine protein ≥ ++ and a confirmed 24-hour urine protein amount> 1.0 g;
* 3. Suffering from active infection, or unexplained fever within 7 days before medication ≥ 38.5℃, or baseline white blood cell count> 15×109/L;
* 4. There are contraindications for immunotherapy (including long-term use of hormones, radiation pneumonia has not been cured and cured within 3 months, etc.);
* 5. Active autoimmune diseases (such as vitiligo, psoriasis, hypothyroidism requiring hormone replacement therapy, etc.);
* 6. Patients with active hepatitis B or C, HIV patients, active tuberculosis, etc.;
* 7. Active infection requires antimicrobial treatment (for example, antibacterial drugs, antiviral drugs, antifungal drugs);
* 8. Known history of allogeneic organ transplantation and history of transplanted hematopoietic stem cells;
* 9. Patients with interstitial lung disease or previous history of interstitial pneumonia;
* 10. Those who have a history of psychotropic substance abuse and are unable to quit or have mental disorders;
* 11. Participated in clinical trials of other anti-tumor drugs within 2 weeks before enrollment;
* 12. Those who have used PD-1/PD-L1 and other immunotherapy drugs before entering the group;
* 13. Previous or concurrently suffering from other uncured malignant tumors, cured skin basal cell carcinoma, cervical carcinoma in situ, and superficial bladder cancer can be included;
* 14. Pregnant or lactating women; those with fertility who are unwilling or unable to take effective contraceptive measures;
* 15. According to the investigator's judgment, there are other factors that may affect the results of the study or lead to the forced termination of the study, such as alcoholism, drug abuse, other serious diseases (including mental illness) need to be treated together, and there are serious laboratory abnormalities , Accompanied by family or social factors, will affect the safety of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
ORR：Objective Response Rate | through study completion, an average of 2 year
  Objective response rate evaluated by Independent Review Committee using radiographic examination according to RECIST1.1

SECONDARY OUTCOMES:
DCR: disease control rate | through study completion, an average of 2 year
  partial rate of subjects evaluated as CR/PR/SD in all subjects
PFS: progression-free survival | through study completion, an average of 2 year
  time from randomization to progression and death
OS: overall survival | through study completion, an average of 2 year
  time from randomization to death

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Province Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided